CLINICAL TRIAL: NCT05497856
Title: Comparison of Integrated Neuromuscular Inhibition Technique With the Myofascial Release on Pain and Stiffness in Rhomboids Trigger Points
Brief Title: Comparison of Integrated Neuromuscular Inhibition Technique With Myofascial Release on Rhomboids Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Naqash Shabbir
Record Dates: First submitted 2022-08-10; First posted 2022-08-11 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: pain pressure threshold; algometer; SPADI
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated neuromuscular inhibition technique (Experimental): ischemic compression, strain counter strain, muscle energy techniques
  Interventions: Other: Integrated neuromuscular inhibition technique
- Myofascial Release (Active Comparator): Deep sustained pressure on the trigger points
  Interventions: Other: Myofascial Release

INTERVENTIONS:
Other: Integrated neuromuscular inhibition technique — Ischemic compression will be applied for 90 seconds followed by the SCS technique with a reduction in pain of at least 70%. it will be held for 20-30 sec followed by the Muscle energy technique in which the isometric contraction will be held for 7-10 sec and then the stretch will be held for 30 sec. This will be repeated 5 times per session with a 30-second rest interval in between each repetition Session will be held 3 times per week for 2 consecutive weeks
  Arms: Integrated neuromuscular inhibition technique
Other: Myofascial Release — Deep sustained pressure on the trigger points will be applied with thumb in 5-7/10 pain tolerance and maintained for 60 seconds and then will be released in a vertical direction followed by stretch of the rhomboid muscle held for 30 sec. This Sustained manual pressure will be applied for 3 times each followed by a stretch per session with a 30 sec rest interval in between .Session will be held 3 times per week for 2 consecutive weeks.
  Arms: Myofascial Release

SUMMARY:
The aim of this research is to compare the effect of integrated neuromuscular inhibition technique and myofascial release on pain, pain pressure threshold and shoulder disability in patients with rhomboid muscle. Randomized controlled trials will be done at Benazir Bhutto Hospital. The sample size is 32. The subjects will be divided in two groups, 16 subjects in integrated neuromuscular inhibition technique group and 16 in myofascial release group. Study duration will be of 6 months. Sampling technique applied will be non-probability purposive sampling technique. Only 25-45 years patients with shoulder/mid back pain and the presence of atleast one trigger point in rhomboid muscles will be included. Tools used in the study are algometer, shoulder pain and disability index (SPADI) and Numeric pain rating scale (NPRS). Data will be analyzed through SPSS 21.

DETAILED DESCRIPTION:
: Trigger points (TrPs) are focal, discrete, and hyperirritable spots located in a taut band within a skeletal muscle. These are painful on compression and can produce referred pain, tenderness, autonomic nervous system symptoms, restricted range of motion and motor dysfunction. These trigger points are developed as a result of trauma, overuse, joint dysfunction, mechanical pressure overload, psychological distress, repetitive overhead activities, and postural stress. Shoulder imbalances can cause tightness of the Rhomboid muscles. The pathogenesis results from the overloading and injury of muscle tissue, leading to involuntary shortening of localized fibers.

However, there is dearth of literature showing the effects of INIT or MFR on trigger points of muscles like Trapezius, IT band, gluteus medius and piriformis etc. Rhomboids trigger points treatment has quiet limited evidence. The available studies focus on these trigger point release by electrotherapy or by muscle energy techniques.

Soft tissue manual mobilization like INIT can provide an effective mean to treat these trigger points as they have beneficial effects in other areas. This study focused on use of both manual techniques to find out their effects on pain, pain pressure threshold and shoulder disability of Rhomboid trigger points. Both manual techniques are easy to administer and require no equipment. INIT is proven to have beneficial effects on multiple muscles of body but its efficacy has not been tested on rhomboid so this study will also add to that and specifically in Pakistan there is no single study has been conducted to compare the effects of INIT and MFR in patients with Rhomboid Trigger Points. The results of this study therefore had therapeutic significance for determining whether the two approaches yield comparable results or whether one is more effective than the other. This would assist in laying the groundwork for more research and developing treatment regimens for the aforementioned population

ELIGIBILITY:
Inclusion Criteria:

* • Shoulder or mid back pain

  * Presence of atleast one trigger points in rhomboids (diagnosed by the characteristics like hyperirritable spot in a taut band, twitch response and referral pain)
  * Presence of Jump sign

Exclusion Criteria:

* • Any history of recent shoulder or Neck surgeries

  * Fractures, Dislocations, Traumatic injuries, Adhesive capsulitis, Tendinitis, thoracic outlet syndrome, Advanced osteoporosis, Psychiatric Disorders
  * Signs of cervical spinal cord compromise (e.g. diffuse sensory abnormality, diffuse weakness, hyperreﬂexia, or the presence of clonus
  * Two or more signs of nerve root involvement (e.g. dermatomal sensation changes, myotomal weakness, or diminished/absent tendon jerk reﬂexes)
  * A history of shoulder degenerative joint disease as per radiographs, endocrine disorders, and autoimmune conditions (e.g. rheumatoid arthritis, ﬁbromyalgia etc)

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
NPRS | 2nd week
  it is a 11 point scale for pain measurements with 0 describing no pain and 10 describing max. pain. changes will be measure from baseline to 2nd week
Pain Pressure threshold | 2nd week
  Pain pressure threshold is measured using algometer. The term algometer may imply pressure tolerance testing, the maximum amount of pressure one may endure. The point at which subjects first said they felt pain was called the Verbal Report of Pain (VRP). The point at which they said the pressure 'hurt a lot' was called the Pain Reaction Point (PRP). changes will be measured from baseline to 2nd week

SECONDARY OUTCOMES:
shoulder pain and disability index (SPADI) | 2nd week
  Shoulder disability will be measured using shoulder pain and disability index (SPADI). The shoulder pain and disability index (SPADI) is a self-report questionnaire developed to measure the pain and disability associated with shoulder pathology. The SPADI consists of 13 items in two subscales: pain (5 items) and disability (8 items). changes will be measured from baseline to 2nd week

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Benazir Bhutto Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No